CLINICAL TRIAL: NCT02594007
Title: Mobile Health Monitoring Solution for Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 774885-1
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Heart Failure
Keywords: telehealth; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- discharge home (Experimental): SEEQ for 28 days. Cardiocom for 30 days
  Interventions: Device: SEEQ; Device: Cardiocom
- discharge to skilled nursing facility (Experimental): SEEQ for 28 days, DocView for 30 days
  Interventions: Device: SEEQ; Device: DocView

INTERVENTIONS:
Device: SEEQ — Mobile cardiac telemetry system worn externally for a total of 28 days.
Device: Cardiocom — Patient-based interface tool that includes a blood pressure cuff and blue-tooth enabled scale for daily recordings. The patient will also answer a series of behavioral and symptomatic questions daily through 30 days.
  Arms: discharge home
Device: DocView — Patient-based interface tool that analyzes state of wellness. The patient will answer a series of questions daily through day 30.
  Arms: discharge to skilled nursing facility

SUMMARY:
Heart Failure (HF) affects 5.7 million Americans and is the only major cardiovascular disorder on the rise. The primary aim of this study is to formally study the combined effects of several different tele-health modalities, all currently approved and available for general use, to determine if such combinations will result in an increase in early intervention and a resultant decrease in acute cardiac decompensation requiring a hospitalization or Emergency Room (ER) visit. This study will attempt to characterize the frequency of health care interventions attributable to the use of these technologies, and any relationship between these interventions and the frequency of hospitalization or ER visits.

Secondary objectives include characterization of healthcare utilization, healthcare costs, and patient experiences with regard to the use the provided technologies.

DETAILED DESCRIPTION:
It is estimated that 400,000 to 700,000 new cases of heart failure (HF) are diagnosed each year and the number of deaths in the United States from this chronic condition has more than doubled since 1979 - averaging 275,000 annually. HF accounts for over 1.1 million annual hospital discharges, 3.4 million physician office visits, 668,000 emergency department visits, and 293,000 outpatient visits per year. The economic impact is equally staggering: the total estimated annual cost of heart failure exceeds $40 billion. This figure is expected to reach $97 billion by 2030. While initial hospitalizations consume a vast amount of health care resources, readmissions are also a significant problem. The overall readmission rate (all cause) in the United States is 19.6%. Studies have shown the 30-day readmission rate for HF to be 24%. The important clinical implication is that patients are particularly vulnerable in the early post-discharge period (30-90 days from hospital to home) and require heightened surveillance, especially if the hospital admission has been prolonged or if the patient has had prior admissions for worsening HF. Despite advances in pharmacologic and monitoring device therapy, the inability to effectively manage and influence patient behavior and the inability of patients to identify signs and symptoms of decompensated HF are major hurdles to improving outcomes and avoiding subsequent readmissions. Less than 10% of HF patients are eligible for implantable monitoring devices due to a variety of reasons. Non-invasive cardiac telemetry units only monitor a patient's echocardiograph (ECG). HF patients present with numerous other physiologic parameters which largely go unmonitored and changes in status undetected after discharge from hospital to home. A worsening status in any one of these indicators may predict worsening condition or decompensation. This gap leaves a tremendous percentage (the majority, in fact) of the HF population at risk for repeat medical crisis and re-hospitalizations.

Managing the HF patient population requires highly skilled clinicians, stringent monitoring and care coordination, and advanced technology integration. The investigators propose a patient-centered non-invasive remote monitoring care system for HF. This model leverages three distinct technology platforms. This unique care plan brings together physiologic data capture with symptomatic and behavioral patient information into a dynamic patient engagement and education mobile platform that analyzes, predicts and notifies clinicians when a patient's baseline health is changing before it leads to a negative health consequence and subsequent hospital re-admission or ER visit.

1. A small cutaneous Mobile Patient Monitoring patch (SEEQ®) from Medtronic that continuously collects ECG data, plus heart rate, heart rate variability, respiratory rate, and atrial fibrillation status. These added physiologic parameters provide clinicians more precise insight into a patient's condition and clearly differentiates the monitoring technology from standard approaches. The Medtronic patch is applied like a band-aid to the patient's chest prior to hospital discharge. As it collects data, the information is wirelessly transmitted via Bluetooth to a patient care platform from which providers can access information in live-time for 30 days post discharge. Medtronic's patch does not require leads like other commercially available systems, and does not need to be removed during bathing and other normal activities. Thus this product increases patient compliance and enhances satisfaction. An increase in patient compliance will ensure a more complete and accurate picture of the patient's health. Captured data is used to 1) provide clinicians with physiological data for patients who are at risk of near-term decompensated HF, and 2) allow clinicians to deliver live-time treatment intervention and guidance from anywhere at any time, preventing health problems from escalating into health crises.

   Another key differentiator in this care model is the patient's use of a tablet-based tele-health mobile software application that includes the patient's discharge plan, a daily medication management list, reminders, and CHAT features for live, interactive communication with the care team. The software assesses the patient's psychosocial status and enables clinicians to coach and guide patients to change negative health behaviors and adhere to their care plan.
2. Medtronic's Cardiocom system deploys a proprietary cellular-based patient interface tool (Commander Flex), a blood pressure cuff that interfaces directly with the Commander Flex and a Bluetooth enabled medical-grade scale that also interfaces directly with the Commander Flex. The patient is required to take the blood pressure and weight measurements at prescribed intervals over the evaluation period (30 days) as well as answer a variety of behavioral and symptomatic questions that operate on a proprietary tree-based questioning algorithm.
3. Docview® mHealth solution encourages self-management and empowers patients to become stakeholders in their health. The application collects real-time data with regular "check-ins" to analyze state of wellness, and enables patients to connect live with their care team - no matter where they are. The entire process takes less than one minute to complete and the answers provide the care team an actionable risk-stratification snapshot. Automating the process allows larger patient populations to be monitored, yet drastically reduces provider-patient involvement, as only at-risk patients need to be notified (10-15% estimated). In a traditional setting, the monitoring team typically calls every patient and could maintain a caseload of only 20-25 patients (average call time 20-25 min). All patients have to be contacted by phone just to determine if a risk exists. The proposed tele-health solution uses real-time data analysis and predictive modeling to proactively notify a provider that a patient's baseline health is changing prior to a negative health issue, and quickly delivers an intervention to the patient based on clinical decisions and statistically validated treatment algorithms.

This unique care plan brings together physiologic data capture with symptomatic and behavioral patient information into a dynamic patient engagement and education mobile platform that analyzes, predicts and notifies clinicians when a patient's baseline health is changing before it leads to a negative health consequence and subsequent hospital re-admission or ER visit.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted patients to Morristown Medical Center located on Gagnon 1 Heart Failure (HF) dedicated unit with an anticipated Discharge DRG of HF
2. Subjects with acute decompensated HF
3. Subject > 55 years of age
4. Subject meets the indications for the use of the external patch
5. Subject is able and willing to provide informed consent

Exclusion Criteria:

1. Subjects with an implantable cardiac device or scheduled to receive a cardiac device within 30 days of enrollment
2. Skilled Nursing Facility (SNF) bound patients who are unwilling/unable to receive care at CareOne Madison
3. Subject with a scheduled readmission within 30 days of discharge
4. Subjects weighing > 500 lbs
5. Subjects with potentially life-threatening arrhythmias, or who require inpatient/hospital monitoring
6. Subject who is expected to receive a heart transplant or a ventricular assist device within 6 months of enrollment
7. Subject with known allergies or hypersensitivities to adhesives or hydrogels
8. Subject who cannot tolerate placement of external patch monitor on chest in the proposed location (electrocardiogram lead II orientation)
9. Subject who will not comply with project protocol requirements (i.e. Docview/Cardiocom engagement). This includes completing required data collection, and attending required follow up visits
10. Prior enrollment in this study
11. Subjects who are pregnant
12. Subjects who are non-English speaking.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12-31 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Hospital readmission or Emergency Room visit | within 30 days of hospital discharge

SECONDARY OUTCOMES:
Clinical interventions initiated by data collected from Cardiocom, SEEQ, and/or Docview | Within 30 days of hospital discharge
  Clinical interventions are defined as any intervention with the participant and may include phone contact, counseling, medication changes, and clinic visits.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Bonnet, APNc MSN RN, Principal Investigator — Morristown Medical Center
Locations (1):
- Morristown Medical Center, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: HFSA 2010 Comprehensive Heart Failure Practice Guideline — http://www.ncbi.nlm.nih.gov/m/pubmed/20610207/